CLINICAL TRIAL: NCT06852274
Title: Management of Symptomatic Uncomplicated Diverticular Disease (SUDD) of the Colon With Clostridium Butyricum CBM588® Versus Rifaximin: Results From a Real-World Retrospective Italian Study
Brief Title: Clostridium Butyricum CBM588® vs. Rifaximin for Symptomatic Uncomplicated Diverticular Disease (SUDD): A Real-World Retrospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Amjad Khan (Other)
Collaborators: San Giovanni Addolorata Hospital (Other)
Responsible Party: Sponsor-Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental medicine, Liaquat University of Medical & Health Sciences
Organization: Liaquat University of Medical & Health Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CESU/104/07.05.2024
Record Dates: First submitted 2025-02-22; First posted 2025-02-28 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Diverticular Diseases; Gastro-Intestinal Disorder
MeSH Terms: conditions — Diverticular Diseases; Digestive System Diseases | interventions — Rifaximin; Tablets

STUDY DESIGN:
Intervention Model Description: This retrospective, real-world clinical study reviewed patient records to evaluate the effectiveness of Clostridium butyricum CBM588® (Butirrisan®) with fiber supplementation for managing Symptomatic Uncomplicated Diverticular Disease (SUDD). Patients who received this probiotic and fiber combination in a routine clinical setting were included. The study assessed symptom reduction, prevention of surgery, and changes in patient-reported outcomes. No prospective randomization was performed, and all data were derived from existing clinical records, reflecting routine clinical practice.
Masking Description: This retrospective, real-world clinical study reviewed patient records to evaluate the effectiveness of Rifaximin with fiber supplementation for managing Symptomatic Uncomplicated Diverticular Disease (SUDD). Patients who received this antibiotic and fiber combination in a routine clinical setting were included. The study assessed symptom reduction, prevention of surgery, and changes in patient-reported outcomes. No prospective randomization was performed, and all data were derived from existing clinical records, reflecting routine clinical practice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic + Fiber Supplementation Group (Probiotic Group) (Other): Participants in this group received Clostridium butyricum CBM588® (Butirrisan®) probiotic at a dose of 3 tablets/day for 1 month, followed by 3 tablets/day for 2 weeks per month for 12 months, in addition to fiber supplementation. These treatments were administered as part of routine clinical care, and data were collected retrospectively from patient records.
  Interventions: Dietary Supplement: Clostridium butyricum CBM588® (Butirrisan®)
- Rifaximin + Fiber Supplementation Group (Control Group) (Other): Participants in this group received Rifaximin 400 mg twice daily for 7-10 days per month along with fiber supplementation. These treatments were administered as part of routine clinical care, and data were collected retrospectively from patient records.
  Interventions: Drug: Rifaximin 400 mg Oral Tablet

INTERVENTIONS:
Dietary Supplement: Clostridium butyricum CBM588® (Butirrisan®) — Probiotic
  Other Names: Butirrisan®, PharmExtracta S.p.A.
  Arms: Probiotic + Fiber Supplementation Group (Probiotic Group)
Drug: Rifaximin 400 mg Oral Tablet — Antibiotic
  Arms: Rifaximin + Fiber Supplementation Group (Control Group)

SUMMARY:
This retrospective, real-world, single-center clinical study aimed to evaluate the effectiveness of probiotic Clostridium butyricum CBM588® (Butirrisan®) versus Rifaximin in the management of Symptomatic Uncomplicated Diverticular Disease (SUDD). Patients with diverticulosis and a history of mild-to-moderate diverticulitis were included, and their clinical outcomes were assessed using existing patient records.

The study compared two treatment groups:

Experimental Group: Clostridium butyricum CBM588® (Butirrisan®) + fiber supplementation.

Control Group: Rifaximin + fiber supplementation.

The primary endpoint was the reduction in SUDD symptoms, evaluated using patient-reported outcomes. Secondary outcomes included assessment of safety, risk of surgery, and changes in abdominal pain frequency and severity.

DETAILED DESCRIPTION:
Diverticulosis is a common condition affecting up to 60% of individuals over 60 years old, with 10-25% developing Symptomatic Uncomplicated Diverticular Disease (SUDD). This condition is characterized by chronic low-grade inflammation, altered gut microbiota, and persistent abdominal symptoms such as bloating, pain, and irregular bowel habits.

Traditional treatment often involves cyclic rifaximin therapy. However, recent studies have highlighted the potential of microbiome-modulating therapies, including probiotics such as Clostridium butyricum CBM588®, to improve gut health, reduce inflammation, and manage SUDD symptoms.

This retrospective, real-world study reviewed clinical records of 70 patients who received treatment for SUDD at a single center. The data were extracted from routine clinical practice records, without any prospective patient recruitment. Patients were categorized into two groups:

The probiotic group received Clostridium butyricum CBM588® (Butirrisan®) with fiber supplementation.

The control group received Rifaximin 400 mg twice daily for 7-10 days per month, alongside fiber supplementation.

Outcomes were measured based on symptom relief over a 12-month period, including the frequency and severity of abdominal pain, the risk of surgery, and patient-reported outcomes. The study provided real-world evidence on the potential benefits of Clostridium butyricum CBM588® in supporting a microbiome-targeted approach for managing SUDD, potentially reducing reliance on antibiotics and improving patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years
* Diagnosed diverticulosis (confirmed by colonoscopy or CT scan)
* History of mild-to-moderate diverticulitis
* Symptomatic Uncomplicated Diverticular Disease (SUDD) requiring management

Exclusion Criteria:

* Prior abdominal surgery
* History of inflammatory bowel disease (IBD) or colorectal cancer
* Use of antibiotics or probiotics within 4 weeks prior to study entry
* Severe chronic comorbidities (e.g., advanced liver or kidney disease)
* Pregnancy or breastfeeding
* Patients with acute diverticulitis within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Symptoms of Diverticular Disease | 12 months
  Assessment Tool: Patient-reported outcome questionnaires derived from clinical records.
  Description: Evaluation of symptom relief, including changes in abdominal pain, bloating, and bowel habit irregularities, based on patient records.

SECONDARY OUTCOMES:
Assessment of Safety and Tolerability of Clostridium butyricum CBM588® | 12 months
  Review of adverse events and overall tolerability of probiotic therapy as documented in clinical records.
Incidence of Surgical Intervention in Patients with Diverticular Disease | 12 months
  Percentage of patients requiring surgical intervention due to complications of diverticular disease, as confirmed by medical records.
  Measurement Tool: Review of surgical records and patient medical charts.
  Unit of Measure: % of patients requiring surgery.
Changes in Abdominal Pain Frequency, Duration, and Severity | 12 months
  Symptom tracking via a validated pain scale extracted from patient records.
  Frequency Scale: 1: <1x/week, 2: 1-2x/week, 3: 3-6x/week, 4: Daily.
  Duration Scale: 1: <30 min, 2: 0.5-1h, 3: 1-6h, 4: >6h.
  Severity Scale: 0: No pain, 1: Mild, 2: Moderate, 3: Severe, 4: Very severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine & Technological Innovation Dept. University of Insubria, Varese, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Urgesi R, Pagnini C, De Angelis F, Khan A, Pallotta L, Fanello G, Antypas P, Di Paolo MC, Villotti G, Bertuccioli A, Sisti D, Di Pierro F, Zerbinati N, Graziani MG. Management of symptomatic uncomplicated diverticular disease (SUDD) of the colon with Clostridium butyricum CBM588 versus rifaximin: a retrospective cross-sectional study. Int J Colorectal Dis. 2025 Oct 18;40(1):216. doi: 10.1007/s00384-025-05005-6. PMID 41108431